CLINICAL TRIAL: NCT06450860
Title: Developing and Testing a Nutrition Support Assessment Tool - An Implementation Trial
Brief Title: Developing a Nutrition Support Assessment Tool
Acronym: NSAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: The MANNA Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: iRISID-2022-1304
Record Dates: First submitted 2024-05-23; First posted 2024-06-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-06

CONDITIONS: Nutrition Assessment; Food Insecurity
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nutrition Intervention (Other): Participants receive an individualized food provision and/or supplemental food support referral based on responses to the NSAT.
  Interventions: Other: Nutrition Interventions

INTERVENTIONS:
Other: Nutrition Interventions — Individualized food provision and/or supplemental referral based on participant's unique needs/responses to assessment (NSAT). Food provision interventions include medically tailored meals, home delivered prepared meals, grocery boxes, grocery delivery services, food pantries, and soup kitchens/meal sites. Supplemental interventions include SNAP benefit enrollment support, nutrition education, and cooking education.

SUMMARY:
The research team developed the Nutrition Support Assessment Tool (NSAT) that incorporates key patient life information (e.g., ability to cook, access to refrigerator/stove, medical conditions and nutritional status) to facilitate individualized nutrition referral. The overall goal of this study is to refine and test the NSAT as a systematic approach to provide individualized nutrition needs screening and referral for patients being discharged from the acute care setting at Jefferson Health. The investigators hypothesize the NSAT will be successful in identifying individualized nutrition referrals that are deemed acceptable and appropriate by enrolled participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Currently admitted to Thomas Jefferson University or Methodist Hospital or Emergency Department
* Has working phone number and is willing to participate in follow-up data collection
* Eats by mouth
* Lives in MANNA's geographic service area
* Patient reports food insecurity or malnutrition using existing screening tools

Exclusion Criteria:

* Unwilling to provide consent
* Unsheltered/unhoused
* Lives in or is being discharged to facility that provides daily meals (e.g., long term care, incarcerated)
* On hospice or has life expectancy of less than 4 months, per clinician
* Not consentable
* Deaf or has other major communication barriers that compromises ability to participate in study activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Reach of Nutrition Interventions | Baseline
  # and type of referrals made based on NSAT results

SECONDARY OUTCOMES:
Uptake of Nutrition Interventions | Week 1 & Week 4
  # and type of referrals accepted and utilized by participants
Acceptability of Nutrition Intervention | Week 1 & Week 4
  Acceptability of nutrition interventions using the Acceptability of Intervention Measure (AIM)
Appropriateness of Nutrition Intervention | Week 1 & Week 4
  Appropriateness of nutrition interventions using the Intervention Appropriateness Measure (IAM)
Satisfaction with Nutrition Intervention | Week 4
  Self-reported satisfaction with nutrition intervention using a research-team developed assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No